CLINICAL TRIAL: NCT04478942
Title: PROMMO Trial: Prelabor Rupture of Membranes Managed With Oral Misoprostol Versus Intravenous Oxytocin
Brief Title: PROMMO Trial: Oral Misoprostol vs IV Oxytocin
Acronym: PROMMO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0770; A532860 (Other: UW Madison); SMPH/OBSTET & GYNECOL (Other: UW Madison); Protocol Version 9/20/2023 (Other: UW Madison); 2020-0240 (Other: UW-Madison IRB)
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Premature Rupture of Membrane; Induction of Labor Affected Fetus / Newborn
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- oral misoprostol (Active Comparator): At time of delivery, participants randomly assigned to either oral misoprostol will receive 50 mcg of Misoprostol every 4 hours up to 6 doses, OR until simplified Bishop score >6 (whichever is achieved first).
  Interventions: Drug: Misoprostol Oral Product
- intravenous oxytocin (Active Comparator): At time of delivery, participants randomly assigned to intravenous oxytocin, will be administered the drug per standard of labor and delivery titrations.
  Interventions: Drug: Intravenous Oxytocin

INTERVENTIONS:
Drug: Misoprostol Oral Product — Misoprostol will be dosed using the preexisting UnityPoint Health-Meriter Protocol for oral misoprostol administration.
  Other Names: Oral Product
  Arms: oral misoprostol
Drug: Intravenous Oxytocin — Intravenous oxytocin administration will also follow standard, UnityPoint Health-Meriter Protocol.
  Other Names: IV Product
  Arms: intravenous oxytocin

SUMMARY:
This is a prospective, randomized trial looking at the ideal method of labor induction for women with prelabor rupture of membranes and an unfavorable cervical Bishop score. The study will compare oral misoprostol and intravenous oxytocin.

DETAILED DESCRIPTION:
The purpose of this study is to look at optimal induction management of prelabor rupture of membranes (PROM) at or beyond 34 weeks gestational age.

Objective 1: To determine if there is a decrease in time from initiation of induction of labor to vaginal delivery in women with an unfavorable cervix with the use of oral misoprostol versus intravenous oxytocin.

Hypothesis: Cervical ripening with misoprostol will be beneficial in women with an unfavorable cervix.

Sub objective 1: To determine if the use of oral misoprostol for cervical ripening decreases the rate of postpartum hemorrhage in women with PROM.

Hypothesis: Misoprostol use will result in significantly lower rate of postpartum hemorrhage.

Sub objective 2: To evaluate the rates of infectious morbidity in peripartum women and neonates exposed to misoprostol versus oxytocin in PROM.

Hypothesis: The use of oral misoprostol will result in lower rates of infectious morbidity in mother and neonate.

Sub objective 3: To analyze patient satisfaction surveys. Hypothesis: Patients in the oral misoprostol group will be more satisfied with their labor experience.

Exploratory Outcome To determine if there is a difference in cost between induction of labor in women with an unfavorable cervix with the use of oral misoprostol versus intravenous oxytocin.

Hypothesis: The use of oral misoprostol will be cost effective in women presenting with PROM and an unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* Early Term to late term pregnancy (>37 weeks and 0 days and <42 weeks and 0 days)
* Late Preterm Pregnancy (34 weeks and 0 days and <37 weeks)
* Confirmed rupture of membranes by either sterile speculum exam or AmniSure
* Simplified Bishop Score ≤ 6
* Maternal Age > 18 years old
* Singleton gestation
* Appropriate gestational age dating by certain LMP or ultrasound performed prior to 20 weeks gestational age

Exclusion Criteria:

* Concern for intra-amniotic infection
* Previous Cesarean delivery
* Lack of appropriate dating criteria for the pregnancy
* Inability to give informed consent in the patient's native language
* Known bleeding disorder such as von Willebrand's disease or hemophilia
* Anticoagulation administration within 24 hours of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Time from initial medication administration to vaginal delivery | Up to 72 hours
  time from initiation of induction of labor to vaginal delivery in women with an unfavorable cervix with the use of oral misoprostol versus intravenous oxytocin

SECONDARY OUTCOMES:
Secondary endpoint 1: Rate of Postpartum Hemorrhage | up to 24 hours for immediate postpartum hemorrhage
  the rate of postpartum hemorrhage in women with prelabor rupture of membranes with use of oral misoprostol for cervical ripening
Secondary endpoint 2: Rate of Suspected or Confirmed Intrapartum Intramniotic Infection | Prior to delivery
  Rates of infectious morbidity in peripartum women and neonates exposed to misoprostol versus oxytocin in prelabor rupture of membranes.
Secondary endpoint 3: Rate of Suspected Endometritis | From delivery to 6 weeks postpartum
  patient satisfaction surveys
Secondary endpoint 4: Rate of Infectious Morbidity for Neonates | up to 6 weeks of life
  Neonatal infection that is diagnosed within the first 6 weeks of life related to maternal infection diagnosed by positive blood cultures or fever.
Secondary endpoint 5: Participant Satisfaction as Measured by modified Labour Agentry Scale | Postpartum day one with repeat instrument at 6 weeks postpartum
  The modified labour agentry scale has scores that indicate satisfaction with the patient's experience in labor

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn Adams, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UnityPoint Health- Meriter Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No